CLINICAL TRIAL: NCT00502346
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled Trial to Determine the Relative Effect of PM101 I.V. Versus Placebo on Hemodynamics in Healthy Adult Volunteers
Brief Title: A Trial to Determine the Relative Effect of PM101 I.V. Versus Placebo on Hemodynamics in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prism Pharmaceuticals (Industry)
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 102
Record Dates: First submitted 2007-07-10; First posted 2007-07-17 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Pharmacodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PM10

SUMMARY:
The primary objective of the study is to compare the effect of PM101 I.V. administered as an immediate intravenous bolus versus placebo on systolic blood pressure. Secondary objectives include evaluation of change from baseline in heart rate and change from baseline to the lowest value in mean arterial pressure and diastolic pressure.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy male or female 18 to 55 years of age, inclusive. Women of childbearing potential must be using a medically acceptable form of birth control for the duration of the trial and must have a negative serum pregnancy test at screening and upon check-in to the study facility.
* Have a BMI within the range of 18-35 kg/m2.
* Be able to communicate effectively with the study personnel.
* Have no significant disease or abnormal laboratory values as determined by medical history, physical examination or laboratory evaluations, conducted at the screening visit or on admission to the clinic.
* Have a normal 12-lead electrocardiogram, without any clinically significant abnormalities of rate, rhythm or conduction (such as high grade AV block, bifascicular or trifascicular block), and a normal QTc interval (i.e., ≤ 450 msec for males and females).
* Be a nonsmoker defined as not having smoked in the past 6 months.
* Be adequately informed of the nature and risks of the study and give written informed consent prior to receiving study medication.

Exclusion Criteria:

* Known hypersensitivity or allergy to amiodarone, Captisol, Cordarone I.V. or its excipients.
* Known hypersensitivity or allergy to iodine or radio-opaque dyes.
* Women who are pregnant or breast feeding.
* A history or presence of asthma or other pulmonary disease, thyroid disease (hypo- or hyperthyroidism), hepatitis or other liver disease.
* Any disease or condition (medical or surgical) which, in the opinion of the investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk.
* The presence of abnormal laboratory values which are considered clinically significant.
* Positive screen for Hepatitis B (HbsAg, Hepatitis B Surface Antigen), Hepatitis C (anti HCV, Hepatitis C Antibody), or HIV (anti-HIV 1/2).
* Received an investigational drug within a period of 30 days prior to enrollment in the study.
* Received any drug therapy within 2 weeks prior to administration of the first dose of any study-related treatment. This exclusion is extended to 4 weeks for any drugs known to induce or inhibit hepatic drug metabolism. However, women of childbearing potential may receive hormonal contraceptives and the investigator may waive short-term use of a medication, which is not specifically prohibited, if the use occurred more than 5 half-lives prior to the first dose of any study-related treatment.
* Consumption of alcohol within 48 hours prior to dose administration or during any in-patient period.
* A positive urine drug screen including ethanol, cocaine, THC, barbiturates, amphetamines, benzodiazepines, and opiates.
* Any history of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction.
* Prior participation in a Prism Pharmaceuticals amiodarone study.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows: 50 mL to 499 mL of whole blood within 30 days, or more than 499 mL of whole blood within 56 days prior to drug administration.
* History of severe respiratory failure, circulatory collapse, severe arterial hypotension, heart failure, cardiomyopathy, or sinus node disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 342 (Estimated)
Dates: Start 2007-07-03 (Actual); Primary Completion 2007-11-02 (Actual); Study Completion 2007-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Anapharm, Montreal, Quebec, Canada